CLINICAL TRIAL: NCT05064514
Title: Single Centre, Prospective, Single Arm Open Label Series of a Transcatheter Tricuspid Valved Stent Graft System for the Reduction of Tricuspid Regurgitation and Improved Patient Reported Outcomes in Patients With Carcinoid Heart Disease
Brief Title: Investigation of a Transcatheter Tricuspid Valved Stent Graft in Patients With Carcinoid Heart Disease
Acronym: TRICAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262072
Record Dates: First submitted 2021-09-16; First posted 2021-10-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Disease; Carcinoid Syndrome; Carcinoid Heart Disease
Keywords: Heart; Valve; Implantation; Transcatheter; Carcinoid
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Serotonin Syndrome; Carcinoid Heart Disease; Carcinoid Tumor

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective single-centre interventional study to test safety and efficacy of the Tricento Transcatheter Tricuspid Valved Stent Graft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter Tricuspid Valved Stent Graft intervention (Experimental): Participants who have carcinoid heart disease with severe symptomatic tricuspid regurgitation and with a significant backflow in the caval and hepatic veins will be treated with the implantation of the Transcatheter Tricuspid Valved Stent Graft
  Interventions: Device: Transcatheter Tricuspid Valved Stent Graft

INTERVENTIONS:
Device: Transcatheter Tricuspid Valved Stent Graft — All participants meeting the inclusion and none of the exclusion criteria will be enrolled. A custom-made Transcatheter Tricuspid Valved Stent Graft based on CT to define anatomic dimensions will be made. The system consists of a custom-made valved stent graft delivery system, a custom-made valved stent graft bioprosthesis and a loading system. The bioprosthesis is self-expanding and consists of a stent graft spanning from the inferior vena cava to the superior vena cava and a lateral bicuspid valve element made of thin porcine pericardial leaflets requiring a low closing pressure, and Nitinol support structures. The participants will undergo a minimally invasive, catheter-based procedure to implant the bioprosthesis which is delivered through a 24 French delivery system via transfemoral access. The device can be repositioned and is retrievable.
  Other Names: TRICENTO

SUMMARY:
The purpose of this investigation is to see if the TRICENTO Valved Stent Graft implant reduces tricuspid regurgitation (TR) and improves the symptoms and quality of life in 15 participants with carcinoid heart disease, and who are not able to have a new valve via a surgical procedure.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks and benefits, participants who provide written consent will be screened to make sure they fulfil the study entry requirements. This will involve a detailed medical history, a CT and an echo scan.

Once it is agreed that the participant is suitable for the study, a custom-made TRICENTO valve is prescribed and made. Participants need to be admitted to hospital for the TRICENTO device to be implanted. Before the device is implanted the participant will have further tests and measurements completed eg ECG, a Cardiac MRI, physical measurements such as height, weight and blood pressure, blood tests, questionnaires and measuring how far they can walk in 6 minutes.

The device is implanted in a cath lab procedure which should take about 30-60 minutes in total. Participants should be discharged from hospital about 2-3 days later after recovery and further echocardiogram, blood tests and questionnaires.

Follow up visits are at 1 month and 6 months after the procedure. The following measurements such as an ECG, echocardiogram, and physical measurements (height, weight and blood pressure), some blood tests, questionnaires and measuring how far they can walk in 6 minutes will be repeated at 1 month and at 6 months after the procedure. A cardiac MRI will also be repeated at 6 months after the procedure. All these tests are to measure whether the TRICENTO valve improves the participant's heart function, symptoms and quality of life.

ELIGIBILITY:
General Inclusion Criteria

* Male or female age ≥18 yrs
* Carcinoid Heart Disease
* NYHA Class II - IV
* Severe symptomatic tricuspid regurgitation
* Inoperable due to active tumour process or patient declines an operative intervention
* Patient willing and able to consent and comply with specified study evaluations
* Adequate understanding of written or spoken English (to complete validated questionnaires)

General Exclusion Criteria

* Previous tricuspid valve repair or replacement
* Permanent vena cava filter
* Mega atrium
* Tricuspid valve stenosis
* Thrombosis of lower venous system
* Severe uncontrolled hypertension (Systolic BP ≥ 180 mmHg and/or Diastolic BP ≥ 110 mm Hg)
* Active endocarditis
* Subject is on chronic dialysis
* Bleeding disorders or hypercoaguable state
* Hemodynamic instability or on IV inotropes
* Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically eg contrast
* Contraindication to anticoagulants or antiplatelet medication
* Known allergy to Nitinol (Titanium or Nickel) alloy, gold or porcine tissue
* Untreated clinically significant coronary artery disease requiring revascularization
* Any Percutaneous Coronary Intervention (PCI) or transcatheter valvular intervention within 30 days prior to the index procedure or planned 3 months post the index procedure
* Myocardial Infarction (MI) or known unstable angina within the 30 days prior to the index procedure
* Pregnant or lactating; or female of childbearing potential with a positive pregnancy test 24 hours before any study-related radiation exposure
* Contraindication to long-term anticoagulation
* Life expectancy according to tumour development is less than 12 months
* Impaired judgment and/or is undergoing emergency treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The number of patients with successful implantation of the TRICENTO bioprosthesis | measured pre intervention and immediately after the intervention
  with a 35% change (reduction) in the V wave pressure in the Inferior Vena Cava (IVC)

SECONDARY OUTCOMES:
To assess the safety of the Tricuspid Valved Stent Graft implantation procedure in patients with carcinoid heart disease with severe symptomatic TR and significant systolic backflow in the hepatic and caval veins, and who are not suitable for surgery. | At baseline, 1 month and 6 months
  * The number of procedural complications (re-interventions related to the device or access procedure, major vascular or bleeding complication (VARC), cardiac death during hospital stay (max 7 days)
  * Rate of death all causes
•To evaluate the reduced symptom burden according to New York Heart Association (NYHA) score | At baseline, and post intervention at 1 month and 6 months
  •NYHA assessment
To evaluate the change in peripheral oedema experienced by patients | At baseline, 1 month and 6 months
  1. measure of ankle circumference (cm)
  2. assessment of oedema scored as: none = 0, ankle = 1, shin = 2, thigh = 3, anasarca = 4
To evaluate the change in of number of admissions to hospital for heart failure | 6 months before procedure and 6 months post implantation.
  Count of number of hospital admissions for heart failure
To evaluate the change in patient reported quality of life (EuroQol- 5 Dimension - EQ5D) | At baseline, and post intervention at 1 month and 6 months
  Measure EQ5D scores for all patients
To evaluate the change in patient reported quality of life (Kansas City Cardiomyopathy Questionnaire (KCCQ)) | At baseline, and post intervention at 1 month and 6 months
  Measure Kansas City Cardiomyopathy Questionnaire scores for all patients
To evaluate the change in patient reported quality of life (Minnesota Living With Heart Failure - MLFHQ) | At baseline, and post intervention at 1 month and 6 months
  Measure MLFHQ scores for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baumbach, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No